CLINICAL TRIAL: NCT03810183
Title: A Multi-center, Proof-of-mechanism Study of Multiple, Oral Doses of Fevipiprant (QAW039) in COPD Patients With Eosinophilia
Brief Title: A Proof-of-mechanism Study of Multiple, Oral Doses of Fevipiprant (QAW039) in COPD Patients With Eosinophilia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAW039E12201; 2018-004267-32 (EudraCT Number)
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: QAW039; Chronic obstructive pulmonary disease; COPD; sputum; eosinophillic; eosinophilia; prostaglandin D2 receptor; DP2; CRTh2; fevipiprant
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Eosinophilia | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This was a subject and investigator-blinded study. Subjects, investigators and all site staff remained blinded to study treatment throughout the study.
  The identity of the treatments was concealed by the use of study drugs that were all identical in packaging, labeling, schedule of administration, appearance, and odor.
  The sponsor could be unblinded to the study treatment at any time, especially in case of a safety concern.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QAW039 450 mg (Experimental): QAW039 (fevipiprant) 450 mg once daily for 6 weeks administered orally as a tablet.
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Placebo once daily for 6 weeks administered orally as a tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — QAW039 (fevipiprant) 450 mg once daily for 6 weeks administered orally as a tablet + Standard of Care
  Arms: QAW039 450 mg
Drug: Placebo — Placebo once daily for 6 weeks administered orally as a tablet + Standard of Care
  Arms: Placebo

SUMMARY:
This was an exploratory, randomized, subject- and investigator-blind, placebo-controlled, parallel group, proof-of-mechanism study of multiple oral doses of fevipiprant (QAW039) in chronic obstructive pulmonary disease (COPD) patients with eosinophilia.

DETAILED DESCRIPTION:
This was an exploratory, randomized, subject- and investigator-blind, placebo-controlled, parallel group, proof-of-mechanism study in COPD subjects with eosinophilia, on standard of care therapy. Standard of care (SoC) treatment in subjects with COPD typically includes a regimen of inhaled corticosteroid (ICS) plus one or more long acting bronchodilator (long-acting beta2-agonist (LABA) or long-acting antimuscarinic antagonist (LAMA)).

The study consisted of a screening period (including an optional pre-screen visit) during which the subject's phenotype and eligibility for the study were assessed. All subjects who met the eligibility criteria after the screening visit were to undergo induction of their sputum to examine the baseline sputum cell counts. Subjects were required to demonstrate both blood and sputum eosinophilia to be eligible for participation in the study.

Eligible subjects were randomized 3:2 to active (fevipiprant 450 mg oral daily) vs. placebo arms. Randomization was stratified by current smoking status (current vs. ex-smoker). Subjects were to continue their COPD standard of care and other medications during the entire course of the study. Subjects were to receive multiple doses of fevipiprant or placebo for six weeks.

Sputum induction was to be repeated at the end of the treatment period and at the end of the study (approximately 4 weeks after the last dose).

The primary purpose of the proof-of-mechanism study was to determine whether fevipiprant (QAW039), when administered to COPD patients with eosinophilic airway inflammation on standard of care therapy, reduced the burden of sputum eosinophilia. Data from other trials did not confirm efficacy of fevipiprant and did not warrant the continuation of treatment in this study. As a result, this study was terminated early.

ELIGIBILITY:
Inclusion Criteria:

1. Acceptable and reproducible spirometry with post-bronchodilator FEV1/FVC < 0.7 and post-bronchodilator FEV1≥ 30 and ≤ 80% of predicted at the screening and baseline visits (GOLD stage II or III COPD).
2. Patients with a physician-diagnosed history of COPD for at least 1 year prior to screening visit, and a documented history of at least one COPD exacerbation within the year prior to screening visit and on a stable therapy regimen for COPD for at least 4 weeks prior to screening visit with inhaled glucocorticoid + one or more long acting bronchodilator.
3. Current or ex-smokers who have a smoking history of at least 10 pack-years (10 pack-years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years, or equivalent).
4. Circulating eosinophils ≥ 300 cells/µL blood AND sputum eosinophils ≥ 3% of total cell count during screening period.

Exclusion Criteria:

1. Patients with a past or current medical history of asthma.
2. Patients with a past or current medical history of conditions other than COPD or allergic rhinitis that could result in elevated sputum eosinophils (e.g., asthma, hypereosinophilic syndrome, Churg-Strauss Syndrome). Patients with known parasitic infestation within 6 months prior to screening are also excluded.
3. Patients who have had a respiratory tract infection or COPD worsening or systemic steroid use within 4 weeks prior to screening visit or between screening and randomization visits.
4. Patients with history of concomitant chronic or severe pulmonary disease (e.g., sarcoidosis, interstitial lung disease, cystic fibrosis, tuberculosis). Exception: patients with concomitant mild or moderate pulmonary hypertension or bronchiectasis are permitted to participate.
5. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective contraception (also called basic contraception)methods during the study.
6. Patients on any statin therapy with a CK level > 2 X ULN at screening.
7. Patients who have a clinically significant laboratory abnormality at the screening visit including (but not limited to):

   * Total white blood cell count <2500 cells/uL
   * AST or ALT > 2.0 X ULN or total bilirubin > 1.3 X ULN
   * Estimated Glomerular Filtration Rate (eGFR) by the Modification of Diet in Renal Disease (MDRD) equation or Bedside Schwartz equation <55 mL/minute/1.73 m2.
8. Patients with any of the following cardiac related concerns:

   * A resting QTcF (Fridericia) ≥450 msec (male) or ≥460 msec (female) at screening visit
   * A history of familial long QT syndrome or known family history of Torsades de Pointe
   * Receiving any medications or other agents known to prolong the QT interval
   * patients with a history of moderate or severe uncontrolled tachyarrhythmias
   * History of a clinically significant cardiovascular event within 1 year prior to the screening visit, such as acute myocardial infarction, congestive heart failure, unstable arrhythmia
   * Patients who, in the judgment of the investigator have a clinically significant ECG abnormality such as (but not limited to) sustained ventricular tachycardia, or clinically significant second or third degree AV block without a pacemaker

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (3):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
- Novartis Investigative Site, Bradford, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 4 investigative sites in 2 countries (Germany and United Kingdom).
Pre-assignment Details: Participants were randomized 3:2 to active (QAW039 450 mg orally daily) vs. placebo arms. Randomization was stratified by current smoking status (current vs. ex-smoker).
Period: Overall Study
Arm/Group | QAW039 450 mg | Placebo
Started | 6 | 3
Completed | 4 | 2
Not Completed | 2 | 1
Not completed — Study terminated by Sponsor | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 450 mg | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (9.71) | 67.3 (6.35) | 64.8 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  White | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Sputum Eosinophil Percentage Based on Log-10 Transformed Scale at Week 6
Description: Sputum eosinophil percentage of the total cell count was obtained from induced sputum samples. Sputum was processed to include preparation of slides for differential cellular count.
  As sputum eosinophil percentage has been found to follow a log-normal distribution, the analysis of this outcome measure was based on log10-transformed scale. The baseline measurement was defined as sputum eosinophil percentage prior to the first dosing (on log10-transformed scale).
Time Frame: Baseline, Week 6
Population: All subjects with available data and no protocol deviations with relevant impact on data.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | QAW039 450 mg | Placebo
Number analyzed (Participants) | 3 | 2
Percentage | -0.43373 (0.39740) | -0.06689 (0.43094)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until last dose plus 30 days, up to a maximum of 72 days.
Description: Any signs or symptoms that occurs during study treatment plus the 30 days post treatment.
Groups:
- QAW039 450mg: QAW039 (fevipiprant) 450 mg once daily for 6 weeks administered orally as a tablet.
- Total: Total
Arm/Group | QAW039 450mg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 4/6 | 2/3 | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 450mg (N=6) | Placebo (N=3) | Total (N=9)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03810183/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT03810183/SAP_001.pdf